CLINICAL TRIAL: NCT05206760
Title: Severe Head Injury Brain Analysis
Acronym: SHIBA
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 271662
Record Dates: First submitted 2021-05-20; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2021-05

CONDITIONS: Brain Injury Traumatic Severe
Keywords: Traumatic Brain Injury; Brain injury classification; Histology
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Brain tissue CSF Blood Urine Saliva Faeces
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trial participants: Patients with severe traumatic brain injury requiring craniotomy or ICP bolt insertion
  Interventions: Procedure: Brain biopsy

INTERVENTIONS:
Procedure: Brain biopsy — Biopsy of brain tissue

SUMMARY:
Safety and feasibility study investigating brain biopsy in severe head injury. When a patient undergoes craniotomy or ICP bolt insertion for trauma, a biopsy of brain tissue is taken.

Blood, saliva, urine and faeces samples are also taken for 7 days following the brain biopsy.

CSF is collected if a CSF drainage device is used.

DETAILED DESCRIPTION:
A minor amendment was submitted to allow histological and immunohistochemical analysis of the samples.

ELIGIBILITY:
Inclusion Criteria: Severe traumatic brain injury -

Exclusion Criteria: Coagulopathy

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have suffered severe traumatic brain injury and require craniotomy or ICP bolt insertion.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-05-16 (Actual); Study Completion 2021-05-16 (Actual)

PRIMARY OUTCOMES:
Feasibility of brain biopsy | immediately after the intervention/procedure/surgery
  Is it feasible to perform brain biopsy through ICP bolt or at time of craniotomy in TBI in order to obtain diagnostic tissue?
Safety of brain biopsy | immediately after the intervention/procedure/surgery
  Is it safe to perform brain biopsy through ICP bolt or at time of craniotomy in TBI?

SECONDARY OUTCOMES:
Classification of TBI | immediately after the intervention/procedure/surgery
  Classify TBI based on histopathological appearances

CONTACTS AND LOCATIONS:
Overall Officials: Chris E Uff, PhD, Principal Investigator — Queen Mary University of London
Locations (1):
- Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers on request. It is anticipated that this pilot study will result in further trials which will have greater data sharing potential.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data are currently available. They will be available for 10 years (until 01/07/2031)
Access Criteria: Apply directly to p.yup@qmul.ac.uk and c.uff@qmul.ac.uk